CLINICAL TRIAL: NCT04009746
Title: Italian Registry of ERCP With Spyglass
Acronym: Spyglass
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: Registro SpyGlass
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Biliary Condition
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) with Spyglass — Endoscopic retrograde cholangiopancreatography (ERCP) with Spyglass

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a procedure used for the diagnosis and treatment of diseases of the biliary tract, pancreas and papilla of Vater. The ERCP allows an indirect vision of the ductal and pancreatic system by means of the endoductal injection of contrast medium and the evaluation of these by X-rays. Recently, cholangioscopy has been developed using the Spy Glass system, introduced on the market in 2007. This allows a direct visualization of the bile duct and pancreatic pathway through the introduction of an optical probe inside the ductal system. SpyGlass was developed to overcome the limitations of traditional cholangioscopy and allow optically guided therapies for the treatment of stenoses and calculations. This is the first cholangioscopy system performed by a single disposable operator (SOC), with two dedicated irrigation channels, an optical channel and a therapeutic channel with a diameter of 1.2 mm. Everything is placed inside a 10 Fr Spy Scope ™ access and delivery catheter (3.3 mm), which allows the tip to flex in 4 directions to facilitate maneuverability and directionality in small ducts.

The irrigation channels of the SOC system allow a fluid flow rate of four to five times higher than that which can be obtained through the operating channel of conventional systems. In bench simulations with loaded Spy Bite ™ biopsy forceps, the SOC system presented a success rate in obtaining access to sites of double interest compared to that of a conventional 2-way limited bending choledocoscope.

Some studies have confirmed the adequacy of the Spy Glass system in providing adequate samples for histological diagnosis and successfully facilitating the treatment of stones.

The new single-use Spy Glass digital display system was introduced in 2014 and no multi-center experience on the use of this device is described to date.

ELIGIBILITY:
Inclusion Criteria:

* With an age above or equal to 18,
* From which informed consent has been obtained,
* Subjected to ERCP carried out by expert operators,
* Subject to ERCP with SpyGlass.

Patients who do not meet all of the listed inclusion criteria will be excluded from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited at the UO of Gastroenterology and digestive endoscopy of the participating centers
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Data collection of characteristics of ERCP with Spyglass | 12 Months
  Frequencies of complications and distribution of population undergoing ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No